CLINICAL TRIAL: NCT04821180
Title: Angle Stable Plate Versus Reverse Shoulder Treatment for Proximal Humeral Fractures: Should the Psychological Health Influence the Choice of Device
Brief Title: Psychological Health Influences the Choice of Device in Proximal Humeral Fractures
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Sponsor
Other Study IDs: HUMERUS-PSY
Record Dates: First submitted 2021-03-22; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Humeral Fracture, Proximal
Keywords: Open reduction and fixation; Reverse shoulder arthroplasty
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients treated by angle stable plate PHILOS
  Interventions: Procedure: Three and four-part proximal humeral fractures' treatment
- patients treated by reverse total shoulder arthroplasty SMR
  Interventions: Procedure: Three and four-part proximal humeral fractures' treatment

INTERVENTIONS:
Procedure: Three and four-part proximal humeral fractures' treatment — Open Reduction and Internal Fixation with angle stable plate PHILOS versus RSA (Reverse Shoulder Arthroplasty

SUMMARY:
It was conducted a prospective study with a series of 63 patients treated with O.R.I.F. (Open Reduction and Internal Fixation) (group A) and with RSA (Reverse Shoulder Arthroplasty) (group B) for three and four-part proximal humeral fractures according to Neer classification system. One independent observer performed clinical and a psychological evaluation at one(T0), six(T1) and twelve months(T2) postoperatively.

The Constant's score and The Disabilities of the Arm, Shoulder and Hand (DASH score) were used for clinical evaluation, while General Anxiety Disorder-7 (GAD-7) and Caregiver Strain Scale (CSS) were used for psychological evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Three and four-part proximal humeral fractures according to Neer classification system;
* Patients seventy years or older;
* Shoulder surgery within one week after trauma

Exclusion Criteria:

* Exposed fractures;
* Pathological fractures;
* Proximal humerus fractures with metaphyseal or diaphyseal extension;
* Contraindications to surgery associated with organ dysfunctions or with coagulopathy;
* Allergy or hypersensitivity to the orthopedic implants;
* Patients who were unable to attend the different follow-ups;
* Patients with psychiatric disorders

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Subjects affected by proximal humeral fractures
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Change in Constant's score | T0 (one-month), T1 (six months), T2 (one year) post operatively
  The shoulder functionality was quantified using the Constant's score ranging between 0 (most disability) and 100 points (least disability).

IPD SHARING:
Plan to Share IPD: No
No sharing